CLINICAL TRIAL: NCT00492947
Title: 0608 GCC:Phase I Study of Intra-tumoral Injection of Dendritic Cells for the Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Dendritic Cell Vaccine for Head and Neck Cancer
Acronym: Dendritic
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: major amendments in progress
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040999
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Phase I; dendritic cell; vaccine; intra tumoral; squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: dendritic cell vaccine — 3 vaccinations total: Day 10, Day 20, Day 30

SUMMARY:
This research study is testing a new treatment of cancer of the head and neck.

Purpose

This research study is being done to:

1. Test the safety of the experimental cancer vaccine made of dendritic cells. An experimental vaccine is one that is not approved by the Food and Drug Administration (FDA).
2. To learn what effects (good and bad) the vaccine will have on you and your head and neck cancer.
3. To learn if the vaccine will stimulate your body's white blood cells, which are part of your immune system (your body's natural defense system).

DETAILED DESCRIPTION:
White blood cells are part of the body's defense system. Sometimes when you have cancer, your body does not know that the cancer cells are making you sick. We hope to teach your white blood cells to find and destroy your cancer cells with a vaccine. The vaccine will be made from a special kind of blood cell called a dendritic cell. This is the cell that will carry the information about your cancer to your white blood cells in your body.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the head and neck in patients with unresectable recurrent disease or distant metastasis or patients who fail conventional radiation therapy and/or chemotherapy and refuse surgical salvage.
* Presence of cervical metastasis that is able to be accessed for injection
* Biopsy accessible tumor (metastatic or primary)
* >18 years of age.
* The following laboratory values obtained ≤14 days prior to registration:

  * ANC ≥1500
  * PLT ≥100,000
  * Hgb ≥ 9.0 g/dL
  * Alkaline phosphatase ≤3 x UNL
  * AST ≤3 x UNL
  * Creatinine ≤1.5 x UNL
* Life expectancy ≥6 months.
* ECOG performance status 0, 1, or 2.
* No chemotherapy for prior 4 weeks.

Exclusion Criteria:

* Pregnant women.
* Nursing women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device {IUD}, abstinence.)
* Known HIV infection.
* Concurrent use of systemic immunosuppressants.
* Other immunocompromising condition that in the opinion of the physician renders the patient a poor candidate for this trial.
* Other active cancer requiring therapy to control the disease.
* Unwillingness to return for follow-up evaluations over a period of up to 2 years following completion of protocol therapy.
* Other intercurrent medical problems that, in the opinion of the investigator, would make participation in the study hazardous for the patient
* Patients in whom the otolaryngologist, radiation oncologist, and medical oncologist can not agree on a consensus node to treat.
* Patients with CNS metastasis or involvement of sites where an inflammatory response would constitute an immediately life threatening situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
safety | 5 years
Efficacy as measured by RECIST criteria | 5 years

SECONDARY OUTCOMES:
Characterize the immune response to the vaccine | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wolf, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Dept. of Otorhinolaryngology, Baltimore, Maryland, United States